CLINICAL TRIAL: NCT01928888
Title: A Randomized, Double-blind, Three-fold Cross-over, Multi-center Study to Compare the Efficacy and Safety of a Single Dose of Oral Talcid (1000 mg Hydrotalcite), a Single Dose of Oral Famotidine 10 mg, and a Single Dose of Placebo in Patients With Acute Heartburn Episodes.
Brief Title: Placebo Controlled Phase IV Study to Compare the Efficacy and Safety of a Single Dose of Oral Talcid, a Single Dose of Oral Famotidine and a Single Dose of Placebo in Patients With Acute Heartburn Episodes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 11201
Record Dates: First submitted 2013-08-20; First posted 2013-08-27 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Heartburn
Keywords: Acute heartburn episodes
MeSH Terms: conditions — Heartburn | interventions — hydrotalcite; Famotidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Arm HFP (Experimental): 1st heartburn episode Intervention Hydrotalcid, 2nd heartburn episode Famotidine, 3rd heartburn episode Placebo
  Interventions: Drug: Talcid (Hydrotalcite, BAY4516H); Drug: Famotidine; Drug: Placebo
- Arm HPF (Experimental): 1st heartburn episode Intervention Hydrotalcid, 2nd heartburn episode Placebo, 3rd heartburn episode Famotidine
  Interventions: Drug: Talcid (Hydrotalcite, BAY4516H); Drug: Famotidine; Drug: Placebo
- Arm FHP (Experimental): 1st heartburn episode Intervention Famotidine, 2nd heartburn episode Hydrotalcid, 3rd heartburn episode Placebo
  Interventions: Drug: Talcid (Hydrotalcite, BAY4516H); Drug: Famotidine; Drug: Placebo
- Arm FPH (Experimental): 1st heartburn episode Intervention Famotidine, 2nd heartburn episode Placebo, 3rd heartburn episode Hydrotalcid
  Interventions: Drug: Talcid (Hydrotalcite, BAY4516H); Drug: Famotidine; Drug: Placebo
- Arm PHF (Experimental): 1st heartburn episode Intervention Placebo, 2nd heartburn episode Hydrotalcid, 3rd heartburn episode Famotidine
  Interventions: Drug: Talcid (Hydrotalcite, BAY4516H); Drug: Famotidine; Drug: Placebo
- Arm PFH (Experimental): 1st heartburn episode Intervention Placebo, 2nd heartburn episode Famotidine, 3rd heartburn episode Hydrotalcid
  Interventions: Drug: Talcid (Hydrotalcite, BAY4516H); Drug: Famotidine; Drug: Placebo

INTERVENTIONS:
Drug: Talcid (Hydrotalcite, BAY4516H) — 2 tablets hydrotalcite (2x500mg) 1000mg and 1 capsule placebo to famotidine
Drug: Famotidine — 2 tablets placebo to hydrotalcite and 1 capsule famotidine 10 mg
Drug: Placebo — 2 tablets placebo to hydrotalcite and 1 capsule placebo to famotidine

SUMMARY:
The purpose of this study is to compare the efficacy and safety of a single oral administration of 1000 mg Talcid® (study medication), a single oral administration of 10 mg famotidine and a single oral administration of placebo (comparator without an active substance) in treating the symptoms of acute heartburn episodes. The study is designed to collect more efficacy data on Talcid® in patients using self-medication to relief the symptoms of acute heartburn.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the age of 18 to 65 years
* A minimum of 6 months history of heartburn
* History of relief of heartburn episodes after self-medication (OTC use) within at least 2 hours
* Occurrence of heartburn episodes at least twice a week during the previous two months
* Severity of heartburn episodes at least 5 on an 11-category heartburn severity scale

Exclusion Criteria:

* History of 'alarming symptoms' e.g. weight loss, vomiting, dysphagia, anemia, hematemesis or melaena
* History of gastric ulcer or gastroesophageal reflux disease requiring regular or intermittent therapy with H2-antagonists or proton pump inhibitors within the previous year
* History of significant gastrointestinal hemorrhage or gastrointestinal surgery
* Gastrointestinal odynophagia (pain during swallowing)
* History or concurrent known duodenitis, pyloric dysfunction with alkaline reflux, motility disturbances, Heliobacter pylori gastritis, or cholelithiasis
* Pregnant or lactating women, or sexually active women of child-bearing potential unless using effective contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 559 (Actual)
Dates: Start 2003-05; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Total heartburn relief over 0-60 min | up to 60 minutes
  The total heartburn relief is claculated as sum of the heartburn relief scores based on a 5-point verbal rating scale.

SECONDARY OUTCOMES:
Total heartburn relief 0-30 min after comparison hydrotalcite vs. placebo and vs famotidine | up to 30 min
  The total heartburn relief is claculated as sum of the heartburn relief scores based on a 5-point verbal rating scale.
Total heartburn relief 0-3 h after comparison hydrotalcite vs. placebo and vs famotidine | up to 3 h
  The total heartburn relief is claculated as sum of the heartburn relief scores based on a 5-point verbal rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (5):
- Germany (5):
  - Frankfurt am Main, Hesse
  - Dresden, Saxony
  - Leipzig, Saxony
  - Berlin, State of Berlin
  - Ask Central Contact